CLINICAL TRIAL: NCT04342663
Title: A Double-blind, Placebo-controlled Clinical Trial of Fluvoxamine for Symptomatic Individuals With COVID-19 Infection
Acronym: STOP COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Eric Lenze, Wallace and Lucille Renard Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202004023
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: COVID 19; Coronavirus
Keywords: COVID 19; fluvoxamine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluvoxamine (Experimental): Start fluvoxamine 100mg capsules, three times daily. May reduce dose (or start at reduced dose) for tolerability reasons. Will be followed in the RCT for approximately 15 days.
  Interventions: Drug: Fluvoxamine
- Placebo (Placebo Comparator): Start placebo one capsule, three times daily. May reduce dose (or start at reduced dose) for tolerability reasons. Will be followed in RCT for approximately 15 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine — Randomized to either fluvoxamine or placebo for approximately 15 days. Will take up to 300mg per day (3 capsules per day) as tolerated.
  Other Names: Luvox
  Arms: Fluvoxamine
Drug: Placebo — Randomized to either fluvoxamine or placebo for approximately 15 days. Will take up to 3 capsules per day as tolerated.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine if a drug called fluvoxamine can be used early in the course of the COVID-19 infection to prevent more serious complications like shortness of breath. Fluvoxamine is an anti-depressant drug approved by the FDA for the treatment of obsessive-compulsive disorder. The use of fluvoxamine for the treatment of COVID-19 is considered investigational, which means the US Food and Drug Administration has not approved it for this use.

This study is fully-remote, which means that there is no face-to-face contact; study materials including study drug will be shipped to participants' houses. Only residents of Missouri and Illinois may participate.

DETAILED DESCRIPTION:
We will consent approximately 152 participants, age 18 and older, who have tested tested positive for COVID-19 and are currently experiencing mild symptoms. All interactions for this study will be conducted remotely by videoconferencing, email, or phone.

Screening: All participants will first complete a pre-screen to see if they may be eligible for the study. Once a participant is confirmed eligible and consented, the study team will send the study materials. These materials will consist of study medication and self-monitoring equipment, including a pregnancy test (for females of childbearing age not using contraception), an oxygen saturation monitor, blood pressure monitor, and thermometer. Once the study team has finalized the screening process, the participant will begin taking the study medication.

RCT: Participants will be randomly assigned (1:1) to take either fluvoxamine or a placebo. This phase of the study will last approximately 15 days and is double-blinded. Participants will take 100mg of fluvoxamine or placebo by mouth three times a day for a daily total of 300mg. They will continue this dose for approximately 15 days. Depending on tolerability, the dose may be adjusted. Participants will also complete short 10-15 minute assessments daily to assess symptoms, results of self-monitoring (including oxygen level, blood pressure, and temperature) and any adverse events.

Open-label Phase: After completing the randomization phase, participants will then participate in an open-label phase (participant will definitely receive fluvoxamine) that will last up to 15 days. Those randomized to placebo will have the opportunity to try fluvoxamine during this time. Those randomized to fluvoxamine will continue this medication while slowly decreasing the drug. The participant may opt out of this phase. The dosage during this time will be 50-100mg two times daily until discontinuing the drug.

Follow-up Phase: We will follow participants for approximately 30 days after the end of the randomized phase. If needed, the study team will review medical records to determine the clinical course of participants.

ELIGIBILITY:
Inclusion Criteria:

1. men and woman age 18 and older;
2. Not hospitalized;
3. Has recently tested SARS-CoV-2 (COVID-19 virus) positive.
4. Currently symptomatic with one or more of one or more of the following symptoms: fever, cough, myalgia, mild dyspnea, diarrhea, vomiting, anosmia (inability to smell), ageusia (inability to taste), sore throat.
5. Able to provide informed consent.

Exclusion Criteria:

1. Illness severe enough to require hospitalization or already meeting study's primary endpoint for clinical worsening.
2. Unstable medical comorbidities including, but not limited to: Severe underlying lung disease (COPD on home oxygen, interstitial lung disease, pulmonary hypertension), decompensated cirrhosis, Congestive heart failure (stage 3 or 4 per patient report and/or medical records).
3. Immunocompromised (solid organ transplant, BMT, AIDS, on biologics and/or high dose steroids (>20mg prednisone per day)
4. Unable to provide informed consent (eg moderate-severe dementia diagnosis)
5. Unable to perform the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - BJC, Belleville, Illinois
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091
- [Derived] Lenze EJ, Mattar C, Zorumski CF, Stevens A, Schweiger J, Nicol GE, Miller JP, Yang L, Yingling M, Avidan MS, Reiersen AM. Fluvoxamine vs Placebo and Clinical Deterioration in Outpatients With Symptomatic COVID-19: A Randomized Clinical Trial. JAMA. 2020 Dec 8;324(22):2292-2300. doi: 10.1001/jama.2020.22760. PMID 33180097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluvoxamine | Placebo
Started | 80 | 72
Completed | 62 | 53
Not Completed | 18 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluvoxamine | Placebo | Total
Number analyzed (Participants) | 80 | 72 | 152
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [35 to 58] | 45 [36 to 54] | 46 [36 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 53 | 109
  Male | 24 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 75 | 66 | 141
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 56 | 50 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Co-existing conditions [Count of Participants; unit: Participants]
  Asthma | 17 | 9 | 26
  Hypertension | 15 | 15 | 30
  Diabetes | 9 | 8 | 17
  High cholesterol | 7 | 7 | 14
  Hyperthyroidism | 6 | 6 | 12
  Anxiety | 5 | 1 | 6
  Arthritis | 4 | 3 | 7
  Depression | 1 | 4 | 5
Body mass index category [Count of Participants; unit: Participants]
  Underweight (<18.5) | 1 | 1 | 2
  Normal (18.5-24.9) | 14 | 7 | 21
  Overweight (25-29.9) | 22 | 22 | 44
  Obese (≥30) | 43 | 42 | 85
Oxygen saturation [Median (Inter-Quartile Range); unit: percentage of oxygen saturation] | 97 [96 to 98] | 97 [96 to 98] | 97 [96 to 98]
Most severe COVID 19 symptom at baseline [Count of Participants; unit: Participants]
  Loss of sense of smell | 26 | 18 | 44
  Fatigue | 17 | 18 | 35
  Body aches | 9 | 13 | 22
  Cough | 9 | 1 | 10
  Subjective fever | 8 | 4 | 12
  Loss of appetite | 3 | 8 | 11
  Chills | 3 | 6 | 9
  Shortness of breath | 2 | 1 | 3
  Loss of taste | 2 | 2 | 4
  Nausea | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Met Clinical Worsening
Description: Clinical worsening is defined meeting both of the following: (1) presence of dyspnea and/or hospitalization for shortness of breath or pneumonia, plus (2) decrease in O2 saturation (<92%) on room air and/or supplemental oxygen requirement in order to keep O2 saturation >92%.
Time Frame: RCT (approximately 15 days)
Population: The primary and secondary end points were measured using participants' self-reported responses on twice-daily surveys during the 15 days after randomization that were corroborated by research staff with phone contact.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 80 | 72
Participants | 0 | 6

2. Secondary Outcome: Clinical Deterioration on a Likert-type Scale (0-6)
Description: (0) none; (1) moderate severity of illness as defined by O2 saturation <92% but no supplemental oxygen requirement; (2) O2 saturation plus supplemental oxygen requirement; (3) O2 saturation <92% plus hospitalization (related to dyspnea/hypoxia); (4) the above, plus ventilator support requirement; (5) the above, plus ventilator support for at least 3 days; (6) death.
Time Frame: RCT (approximately 15 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 80 | 72
Participants
  0 (none) | 80 | 66
  1, shortness of breath and oxygen saturation less than 92% but no supplemental oxygen needed | 0 | 2
  2, O2 saturation plus supplemental oxygen requirement | 0 | 0
  3, oxygen saturation less than 92% + supplemental O2 and hospitalized related to dyspnea or hypoxia | 0 | 3
  4, the above, plus ventilator support requirement; | 0 | 0
  5, oxygen < 92%, + supplemental O2, hospitalized related to dyspnea/hypoxia + ventilator 3 days | 0 | 1
  6, Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected daily via participant self-report during the 15 day RCT and again at the 30 day follow-up for both the fluvoxamine and placebo groups.
Arm/Group | Fluvoxamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/72
Serious Adverse Events (participants affected / at risk) | 1/80 | 6/72
Other Adverse Events (participants affected / at risk) | 13/80 | 28/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluvoxamine (N=80) | Placebo (N=72)
Dehydration (General disorders) | 1 (1) | 0 (0)
Exacerbation of COVID 19 with hospitalization (General disorders) | 0 (0) | 1 (1) — Hospitalized for nausea, vomiting, and chest pain (O2 not below 92%)
Flank Pain (hospitalized) (General disorders) | 0 (0) | 1 (1)
Exacerbation of COVID 19 with hospitalization (General disorders) | 0 (0) | 1 (1) — Hospitalized for nausea, vomiting, fever, low oxygen saturation, and pneumonia
Acute chronic respiratory failure with hypoxia and hypercapnia (hospitalized) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bilateral multi-focal pneumonia with shortness of breath and low oxygen saturation (hospitalized) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Exacerbation of COVID 19 with hospitalization (General disorders) | 0 (0) | 1 (1) — Hospitalized with nausea, fever, and pneumonia with requirement of supplemental oxygen to maintain oxygen saturation about 92%
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluvoxamine (N=80) | Placebo (N=72)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Headache or head pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroenteritis, nausea, or vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacterial infection (General disorders) | 1 (1) | 0 (0)
Vasovagal syncope (General disorders) | 1 (1) | 0 (0)
Teeth chattering (General disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Low oxygen saturation or hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Chest pain or tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Flank pain (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
It was a small study and was conducted within a single geographic area; there was a small number of end point events; it is possible that the differences in clinical deterioration may have been a reflection of the comparative baseline distributions of O2 saturation rather than an effect of treatment; the method of measuring the most severe baseline symptom over time did not appear to provide valid data; the follow-up was short; the 7-point scale created for this study has not been validated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT04342663/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT04342663/ICF_001.pdf